CLINICAL TRIAL: NCT06244212
Title: Topical Treatment for Atopic Dermatitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00108458
Record Dates: First submitted 2024-01-29; First posted 2024-02-06 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Atopic Dermatitis
Keywords: Medication adherence; topical medications; Triamcinolone
MeSH Terms: conditions — Dermatitis, Atopic; Medication Adherence | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Adult or pediatric patients with active dermatitis who receive dermatologic care at Atrium Health Wake Forest Baptist, Department of Dermatology.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Demonstration (Active Comparator): Observe a live demonstration instructing how to dispense 1 fingertip unit (FTU) of medication (triamcinolone cream) per 1% body surface area
  Interventions: Other: Demonstration of applying triamcinolone cream
- Mobile Application (Experimental): Additional mobile application that provides instructions to apply the medication (triamcinolone cream)
  Interventions: Behavioral: Mobile App Use
- Written/verbal instructions only (Other): Standard of care written/verbal instructions only
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Demonstration of applying triamcinolone cream — Live demonstration of applying 1 fingertip unit of triamcinolone cream
  Arms: Demonstration
Behavioral: Mobile App Use — Additional mobile application that provides amount dispensed and adherence data.
  Arms: Mobile Application
Other: Standard of Care — Written/verbal instructions only
  Arms: Written/verbal instructions only

SUMMARY:
Medication adherence is a poorly studied phenomenon that challenges both patients and physicians. 50% of individuals with chronic disease are not adherent to their medication regimen. Within the United States, non-adherence to medical treatment leads to approximately $100 billion in hospital admission costs. While the issue of adherence is not limited to any particular field of medicine, non-adherence occurs in approximately one-third to one-half of dermatological patients. Non-adherence is of importance as it is a significant cause of treatment failure, resulting in worse quality of life, worse health outcomes, and increased insurance costs.

DETAILED DESCRIPTION:
Unlike most modes of medication administration, topical medications do not have a standardized method of dosage administration] Although qualitative administration measures exist, these measures are often arbitrary and not quantifiable (i.e., "a fingertip"). In such cases, inappropriate dosing (i.e., using too much or too little) is an essential cause of treatment failure, and measurements of adherence for topical medications should consider the amount of medication administered. In a study analyzing the response to treatment in psoriatic patients, patients who received a standardized dose of topical calcipotriol achieved a more significant decrease in mean Psoriasis Area and Severity Index (PASI) (47%) compared to patients who were not standardized (17%, P<0.0001). Moreover, over two-thirds of psoriatic patients deemed initially poor responders in the standardized regimen group were considered responsive to treatment after further consideration.

Given topical options' low cost, efficacy, and excellent safety profiles, they are the first line treatment option for mild-to-moderate Atopic Dermatitis (AD) treatment. This study will aim to assess differences in the amount of medication dispensed in two groups of patients with atopic dermatitis. The first will undergo a brief educational demonstration by a trained professional to highlight the appropriate amount of topical medication to dispense for their disease involvement. The second group will be a control group and receive the same medication; however, the Participants will receive standard of care education (verbal and written instructions) only. Data from the two groups will be collected and analyzed to measure trends in dosing (i.e., if the correct dosage quantity and frequency was dispensed).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of skin dermatitis
* Age > 9
* Ability to return for a one-week clinical studies follow-up
* Patients who are candidates for treatment with 0.1% triamcinolone ointment (even if they weren't in the study)
* Adult or pediatric patients with active dermatitis who receive dermatologic care at Atrium Health Wake Forest Baptist, Department of Dermatology.

Exclusion Criteria:

* Patients without the diagnosis of skin dermatitis
* Inability to return for a one week follow up appointment
* Body Surface Area (BSA) affected <2%

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-09-19 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Amount of Topical Medication Dispensed - Demonstration Group | Day 7
  Amount of Topical Medication Dispensed in grams
Amount of Topical Medication Dispensed - Standard of Care Group | Day 7
  Amount of Topical Medication Dispensed in grams
Amount of Topical Medication Dispensed - Mobile Application Group | Day 7
  Amount of Topical Medication Dispensed in grams
Number of times of Application - Demonstration Group | Day 7
  Frequency of Application
Number of times of Application - Standard of Care Group | Day 7
  Frequency of Application
Number of times of Application - Mobile Application Group | Day 7
  Frequency of Application
Change in Investigator Global Assessment (IGA) Scores | Baseline and Day 7
  The IGA is a five-point scale that provides a global clinical assessment of AD severity ranging from 0 to 4, where 0 indicates clear, 2 is mild, 3 is moderate, and 4 indicates severe AD. A decrease in score relates to an improvement in signs and symptoms.
Change in Percentage of Body Surface Area (BSA) affected | Baseline and Day 7
  Body Surface Area percentage = 0.007184 x (Height(cm)^0.725) x (Weight(kg)^0.425)
Subject Questionnaire Scores | Day 7
  a brief questionnaire will be distributed to gain insight into attitudes towards medication samples and educational demonstrations.

CONTACTS AND LOCATIONS:
Overall Officials: Steven R Feldman, MD, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No